CLINICAL TRIAL: NCT01895322
Title: A Phase 2, Multi-center, Open-label, Dose-finding Trial to Investigate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of OPC-41061 in Patients With Chronic Renal Failure Undergoing Peritoneal Dialysis
Brief Title: Open-label Dose-finding Trial of OPC-41061 in Patients With Chronic Renal Failure Undergoing Peritoneal Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-12-002; JapicCTI-132181 (Other: Japan Pharmaceutical Information Center)
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Renal Failure
Keywords: Tolvaptan; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-41061 (Experimental)
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061

SUMMARY:
To investigate the efficacy, pharmacokinetics, pharmacodynamics, and safety of OPC-41061 in patients with chronic renal failure who are undergoing peritoneal dialysis, using daily urine volume, body weight, and edematous conditions as parameters and conducting dose escalation every 2 days until reaching the dose that achieves urine volume increase and then performing 5-day repeated administration at the fixed dose, the final dose used in the dose escalation period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic renal failure
* Patients who are undergoing peritoneal dialysis (continuous ambulatory peritoneal dialysis [CAPD])
* Patients who, after undergoing peritoneal dialysis, received any of the following medical treatments for fluid overload [OR: hypervolemia] that had insufficient effect:

  * Addition or increase of diuretics
  * Increase in concentration or volume of peritoneal dialysis fluid
  * Increase in the number of changes of peritoneal dialysis fluid
* Subjects who, together with their partner, are able to practice one of the specified contraceptive methods until 4 weeks after the final trial drug administration
* Subjects who are inpatients or who can be admitted to the trial site for the duration of the trial period

Exclusion Criteria:

* Subjects with any of the following diseases, complications, or symptoms:

  * Suspected hypovolemia
  * Daily urine volume less than 200 mL
  * Urination impaired due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
  * Cardiac function of NYHA class 4
* Subjects with any of the following medical histories:

  * History of cerebrovascular disorder or coronary artery disease within 4 weeks prior to informed consent
  * History of hypersensitivity or idiosyncratic reaction to benzazepine derivatives such as mozavaptan hydrochloride or benazepril hydrochloride
* Subjects with any of the following abnormal laboratory values:

Hemoglobin lower than 9.0 g/dL, total bilirubin higher than 3.0 g/dL, ALT (GPT) or AST (GOT) 2 times the upper limit of the reference range of the trial site, serum sodium higher than the upper limit of the reference range of the trial site, serum sodium lower than 125 mEq/L, or serum potassium higher than 5.5 mEq/L

* Subjects with any of the following conditions, concomitant diseases, or symptoms:

  * defect in diaphragm
  * hemorrhagic diathesis due to uremia
  * suspected lactic acid metabolic disorder
  * suspected peritonitis, peritoneal damage, peritoneal adhesion, or disorders in intraabdominal organs
* Subjects who have undergone peritoneal dialysis for 8 years or longer
* Subjects who are scheduled to undergo hemodialysis or concomitant use of hemodialysis, or renal transplantation
* Subjects who have participated in any other clinical trial or post-marketing clinical studies within 30 days prior to informed consent
* Subjects who have previously received OPC-41061
* Subjects who are unable to sense thirst or who have difficulty with fluid or food intake
* Female subjects who are pregnant, possibly pregnant, or nursing, or who plan to become pregnant during the trial period
* Subjects otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (6):
- Japan (6):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-41061: In the dose-escalation period,the dose of OPC-41061 was to be sequentially increased every 2 days as indicated below until daily urine volume of the OPC-41061 administration at each dose showed an crease of at least 500 mL from the pre-observation period. Dose escalation was to be terminated at the dose at which daily urine volume increased by 500 mL or more. If an increase in daily urine volume of at least 500 mL was not observed at the dose of 60 mg/day, the subject was to be withdrawn from the trial.
  - 7.5, 15, 30, 60 mg/day (up to a total of 8 days)
  OPC-41061 was administered at a fixed dose (final dose administered in the dose-escalation period) once daily for 5 days on the repeated-administration period.
Period: Overall Study
Arm/Group | OPC-41061
Started | 20
Completed | 7
Not Completed | 13
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 10

BASELINE CHARACTERISTICS:
Arm/Group | OPC-41061
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  Japan | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Urine Volume From Baseline
Description: Change in daily urine volume from baseline during the repeated-administration period (For five days).
Time Frame: Urine Volume on day13 minus Urine Volume at baseline(day9) on the repeated-administration period.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OPC-41061
Number analyzed (Participants) | 7
mL | 18.3 (340.2)

2. Secondary Outcome: Change in Body Weight From Baseline
Description: Change in body weight from baseline during the repeated-administration period(For five days).
Time Frame: Body weight on day13 minus Body weight at baseline(day9) on the repeated-administration period
Measure: Mean (Standard Deviation); unit: kg
Groups:
- OPC-41061: In the dose-escalation period,the dose of OPC-41061 was to be sequentially increased every 2 days as indicated below until daily urine volume of the OPC-41061 administration at each dose showed an increase of at least 500 mL from the pre-observation period. Dose escalation was to be terminated at the dose at which daily urine volume increased by 500 mL or more. If an increase in daily urine volume of at least 500 mL was not observed at the dose of 60 mg/day, the subject was to be withdrawn from the trial.
  - 7.5, 15, 30, 60 mg/day (up to a total of 8 days)
  OPC-41061 was administered at a fixed dose (final dose administered in the dose-escalation period) once daily for 5 days on the repeated-administration period.
Arm/Group | OPC-41061
Number analyzed (Participants) | 7
kg | -0.61 (0.84)

3. Primary Outcome: Percent Change in Daily Urine Volume From Baseline
Description: Percent change in daily urine volume from baseline during the repeated-administration period (For five days).
Time Frame: 100%*<Urine Volume on day13 minus Urine Volume at baseline(day9) on the repeated-administration period/Urine Volume at baseline(day9) on the repeated-administration period>
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | OPC-41061
Number analyzed (Participants) | 7
Percentage | 8.89 (33.2)

4. Secondary Outcome: Percent Change in Body Weight
Description: Percent change in body weight from baseline during the repeated-administration period(For five days).
Time Frame: 100%*<Body weight on day13 minus Body weight at baseline (day9)/Body weight at baseline(day9)>
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | OPC-41061
Number analyzed (Participants) | 7
Percentage | -0.92 (1.31)

ADVERSE EVENTS:
Time Frame: daily for 13 days
Groups:
- OPC-41061: OPC-41061
Arm/Group | OPC-41061
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-41061 (N=20)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Thirst (General disorders) | 3 (3) — General disorders and administration site conditions
Nasopharyngitis (Infections and infestations) | 2 (2)
Blood sodium decreased (Investigations) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No